CLINICAL TRIAL: NCT02491216
Title: A Study on Effects of Acupressure Among the Frail Elderly in Homes for the Aged and Care and Attention Homes for the Elderly
Brief Title: A Study on Effects of Acupressure Among the Frail Elderly in Residential Care Services for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Yan Chai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTC1215-2
Record Dates: First submitted 2015-06-11; First posted 2015-07-07 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Impaired
Keywords: Frailty; Frail elderly; Acupressure; Pragmatic Randomised Controlled Trial
MeSH Terms: conditions — Frailty | interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupressure Group (Experimental): A 15 minutes structured acupressure protocol with specific acupoints and applications technique will be performed on the elderly participants twice a week by the research team in YCHSS Homes. Designated para-medical staffs working in the elderly home or informal care giver of the elderly will be trained and perform the same acupressure protocol on the elderly at 2 additional occasions during the week. The total trial period is 12 weeks.
  Interventions: Other: Acupressure
- Control Group (No Intervention): No acupressure therapy will be provided during the study.

INTERVENTIONS:
Other: Acupressure — A 15 minutes structured acupressure protocol with specific acupoints and applications technique will be performed on the elderly participants twice a week by the research team in YCHSS Homes. Designated para-medical staffs working in the elderly home or informal care giver of the elderly will be trained and perform the same acupressure protocol on the elderly at 2 additional occasions during the week. The total trial period is 12 weeks.
  Other Names: Tui-na
  Arms: Acupressure Group

SUMMARY:
Acupressure has been used for thousands of years in China. Through applying pressure on the specific acupoints based on Traditional Chinese Medicine theory, acupressure could promote relaxation and wellness, balance yin-yang and treat diseases.

The PI has been using acupressure to treat various diseases in the clinics of the School of Chinese Medicine, The University of Hong Kong. Acupressure has demonstrated significant efficacy in treating geriatric diseases, obstetric diseases, pediatric diseases, rheumatoid arthritis and various painful symptoms. When applying acupressure on the Head- Neck - Shoulder area, it could also help to improve insomnia, reduce pain, and regulate the mood of the patients.

"Frailty" is a geriatric syndrome of growing importance in the medical field. Prevalence of frailty increases with age. As our life expectancy increase, there will be more elderly suffered from frailty in the later stage of their life. Although there is still a lack of universally accepted clinical definition for frailty, the syndrome is now commonly understood as decreased reserves in multiple systems, and lowered resilience to negative stress. Frailty could be initiated by single or multiple conditions including malnutrition, chronic diseases, lack of exercise, stress and physiological or social changes caused by aging. Its manifestation includes sarcopenia, anorexia, energy reduction, dysfunctional neuroendocrine system and a pro-inflammatory state. Frailty could affect the emotional state of the elderly, meanwhile, positive affect is protective against the functional and physical decline associated with frailty. There is limited treatment or medication for frailty. The investigators believe that acupressure could be a possible non invasive means to improve the general health conditions, including the emotional conditions of the frail elderly. In the past 2 years, the school of Chinese Medicine has been promoting acupressure as a health maintenance technique to the elderly, mostly frail elderly living in the community dwelling through seminars. It is in investigator's interest to run a prospective research to further understand the efficacy of acupressure in a wider range of frail elderly. The investigators would like to use a well-designed pragmatic randomized controlled trial (PRCT) to investigate if acupressure could help the frail elderly to improve their general quality of life

DETAILED DESCRIPTION:
The research is a collaborative project by The University of Hong Kong and Yan Chai Hospital, with the aim of investigating the potential benefits of applying acupressure regularly on frail elderly. The study is designed as a prospective randomized control trial with the primary objective to investigate if acupressure could help the elderlies to improve their general quality of life.

"Frailty" is a geriatric syndrome of growing importance in the medical field. Although there is still a lack of universally accepted clinical definition for frailty, the syndrome is now commonly understood as decreased reserves in multiple systems, and lowered resilience to negative stress. Frailty could affect the emotional state of the elderlies; meanwhile, positive affect is protective against the functional and physical decline associated with frailty. Since there is limited treatment or medication for frailty. The investigators would like to investigate if acupressure could be a possible non-invasive means to improve the general health conditions, including the psycho-social well being of the frail elderly.

The aim of this research is to study potential beneficial effects of acupressure on a group of frail elderly living in the Homes for the Aged and Care and Attention Homes for the Elderly.

In this study, the investigators will use Tilburg Frailty Indicator (TFI) to assess the frailty level of the elderly.

I. Trial Design:

This is a multicenter, pragmatic randomized control trial (PRCT) with a prospective design.

Hypothesis:

1. Applying regular acupressure (4 times a week, totally 12 weeks) on frail elderly in residential care will improve one or more of the following aspects:

   * Elderly's quality of life
   * Elderly's sleeping quality
   * Elderly's Blood pressure/heart rate
2. Regular acupressure provides additional benefit to the frail elderly in residential care on top of their regular exercise program 108 frail elderlies currently served by the Homes for the Aged and Care and Attention Homes for the Elderly of the Yan Chai Hospital, Social Services Department (YCHSS) will be recruited. All these elderlies are currently participating in the exercise program offered by the residential services of YCHSS. All applications will be screened by the para-medical staffs in the residential services based on the inclusion and exclusion criteria. Qualified applicants will be invited for a health assessment conducted by registered Traditional Chinese Medicine practitioner in the research team to confirm their suitability and invite them to sign the consent form. The consented elderlies will be allocated randomly into treatment group and control group. Randomization is done by computer generated number list in block of 4.

II. Intervention The enrolled elderly will participate in all the assessments and continue to participate in the exercise program offered by the residential care of YCHSS.

Acupressure Group:

A 15 minutes structured acupressure protocol with specific acupoints and applications technique will be performed on the elderly participants twice a week by the research team in YCHSS Homes. Designated para-medical staffs working in the elderly home or informal care giver of the elderly will be trained and perform the same acupressure protocol on the elderly at 2 additional occasions during the week. The total trial period is 12 weeks.

The acupressure treatment involved 12 steps, and mainly concentrates on the acupoints on face, head, neck and shoulder. The treatment is designed to be operated by layman. The acupoints chosen are all easy to be located. All the movements/steps selected are well established and commonly used in the Traditional Chinese Medicine practices. Any movement that demand professional training or involve potential risk (e.g. joint mobilization) is excluded from the protocol. The total treatment process will last for approximately 15 mins.

All the elderly will be invited to participate in a lecture of health care in Chinese medicine after the research.

Control group:

No acupressure therapy will be provided during the study. All the elderly will be invited to participate in a lecture of health care in Chinese medicine after the research.

III. Assessment of Efficacy Efficacy of the treatments will be measured in multi dimensions before and after the treatment for both groups. Time Frame of the assessment are: (1) Baseline; (2) Change from baseline after 12 weeks; (3) Change from baseline at 6th month. The primary outcomes will be the change in quality of life of the frail elderly. The secondary outcomes will be sleeping quality and physiological aspects of the frail elderly. All instruments employed are international recognized and provide an absolute score in measurement.

ELIGIBILITY:
Inclusion Criteria:

* a. Age: 65 years and older;
* b. Gender: male or female;
* c. Currently is a client served by the Residential Care services of YCHSS;
* d. Demonstrate frailty: score 5 or more in the Tilburg Frailty Indicator (TFI);
* e. Physically fit to sit on a normal chair for 15-20 mins for acupressure treatment;
* f. Cognitively competent to understand the instruction from the practitioner and participate actively in the exercise program offered by the Residential Care of YCHSS);
* g. Cognitively competent to sign the consent form: score 6 or more in Abbreviated Mental Test (AMT, Hong Kong Version);
* h. Signed the Patient/Subject Consent Form for this study.

Exclusion Criteria:

* a. Who is currently receiving acupressure or acupuncture as a regular therapy;
* b. Who is decision impaired and unfit to sign the consent form;
* c. Who is suffering from one of the related contraindications for acupressure (including open sores; undiagnosed rashes; high fever; hypertensive emergence; sore and enlarged lymph nodes; the site of an injury, surgery or injection; burn wounds; skin ulcers and eczema);
* d. Who is unable to comply to the set treatment schedule (20% non compliance is allowed).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change of quality of life | Baseline, 12 weeks, 6th months
  questionnaire: Short Form 12 questions Health Survey version 2 (SF-12,v2), Version for Hong Kong Chinese will be used to measure the quality of life of the elderly pre-treatment and post treatment.

SECONDARY OUTCOMES:
change of sleeping quality | Baseline, 12 weeks, 6th months
  questionnaire: Pittsburgh Sleep Quality Index (PSQI) will be used to assess the change in sleeping quality of the frail elderly pre-treatment and post treatment.
change of blood pressure | Baseline, 12 weeks, 6th months
  Sphygmomanometer：Record of the blood pressure of the frail elderly will be logged pre- treatment and during the 12 weeks treatment period on a weekly basis.
change of heart rate | Baseline, 12 weeks, 6th months
  Sphygmomanometer：Record of the heart rate of the frail elderly will be logged pre- treatment and during the 12 weeks treatment period on a weekly basis.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Chinese Medicine, The University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee EJ, Frazier SK. The efficacy of acupressure for symptom management: a systematic review. J Pain Symptom Manage. 2011 Oct;42(4):589-603. doi: 10.1016/j.jpainsymman.2011.01.007. Epub 2011 Apr 30. PMID 21531533
- [Background] Department of Economic and Social Affairs Population Division, United Nations. World Population Aging: 1950-2050. United Nation Publication, 2001.
- [Background] Ostir GV, Ottenbacher KJ, Markides KS. Onset of frailty in older adults and the protective role of positive affect. Psychol Aging. 2004 Sep;19(3):402-8. doi: 10.1037/0882-7974.19.3.402. PMID 15382991
- [Background] Gobbens RJ, van Assen MA, Luijkx KG, Wijnen-Sponselee MT, Schols JM. The Tilburg Frailty Indicator: psychometric properties. J Am Med Dir Assoc. 2010 Jun;11(5):344-55. doi: 10.1016/j.jamda.2009.11.003. Epub 2010 May 8. PMID 20511102
- [Background] Pialoux T, Goyard J, Lesourd B. Screening tools for frailty in primary health care: a systematic review. Geriatr Gerontol Int. 2012 Apr;12(2):189-97. doi: 10.1111/j.1447-0594.2011.00797.x. Epub 2012 Jan 10. PMID 22233158
- [Background] Chu LW, Pei CKW, HoMH et al. Validation of the Abbreviated Mental Test (Hong Kong version) in the elderly medical patient. Hong Kong Med J 1995;1:207-211.
- [Background] Lam CL, Tse EY, Gandek B. Is the standard SF-12 health survey valid and equivalent for a Chinese population? Qual Life Res. 2005 Mar;14(2):539-47. doi: 10.1007/s11136-004-0704-3. PMID 15892443
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- See also: The International Quality of Life Assessment (IQOLA) Project, which is in its tenth year, is translating, validating, and norming the SF-36 Health Survey for use in multinational clinical trials and other international studies. — http://www.iqola.org/countries.aspx